CLINICAL TRIAL: NCT04014205
Title: A Phase I/II，Multicenter, Open-Label, Study of a Novel Bruton's Tyrosine Kinase Inhibitor, Orelabrutinib, in Patients With B-Cell Malignancies
Brief Title: A Study of Tyrosine Kinase Inhibitor Orelabrutinib (ICP-022) in Patients With r/r B-Cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00107
Record Dates: First submitted 2019-06-18; First posted 2019-07-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Part 1：r/r B-cell Malignancies; Part 2：B-cell Malignancies
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Dose Escalation (Experimental): Patients with r/r B-cell malignancies including Grades 1-3a FL, MZL, MCL, and CLL/SLL
  Interventions: Drug: Orelabrutinib (ICP-022)
- Part 2 Dose Expansion (Experimental): Arm 1: Patients with r/r MCL
  Arm 2: Patients with other types of B-cell malignancies, including:
  * CLL/SLL with/without prior treatment
  * r/r FL
  * r/r MZL
  Interventions: Drug: Orelabrutinib (ICP-022)

INTERVENTIONS:
Drug: Orelabrutinib (ICP-022) — ICP-022 The drug product is a white, round, uncoated tablet

SUMMARY:
This is a Phase I/II, multicenter, open-label study to evaluate the safety, efficacy, tolerability, and pharmacokinetics of a novel BTK inhibitor, Orelabrutinib (ICP-022) in Patients with B-cell malignancies. The study contains two parts, Part 1 (dose escalation) and Part 2 (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent.
2. Age ≥ 18 years.
3. Part 1: Patients with histologically confirmed relapsed or refractory B-cell malignancies, including Grades 1-3a FL, MZL, MCL, and CLL/SLL.

   Part 2: Patients with histologically confirmed B-cell malignancies including r/r FL, r/r MZL and CLL/SLL with/without prior treatment.
4. Life expectancy (in the opinion of the investigator) of ≥ 4 months.
5. ECOG performance status of 0 ~1.
6. Must have adequate organ function.
7. Negative test results for HBV ([HBsAg (-)] and non-active HBV or HCV infection

Exclusion Criteria:

1. Pregnant or breast-feeding or intending to become pregnant during the study.
2. Prior treatment with systemic immunotherapeutic agents.
3. Known allergies to Orelabrutinib (ICP-022) or its excipients or infection with HIV.
4. Treatment with any chemotherapeutic agent, or any other investigational therapies within 4 weeks prior to first dose of the study drug.
5. History of allogeneic stem-cell (or other organ) transplantation or confirmed progressive PML.
6. Any external beam radiation therapy within 6 weeks prior to the first dose of the study drug.
7. Concurrent use of warfarin or other vitamin K antagonists or anticoagulation therapies or strong CYP3A inhibitor.
8. Active uncontrolled infections.
9. Recent infection requiring IV anti-infective treatment that was completed ≤ 14 days before the first dose of study drug.
10. Unresolved toxicities from prior anti-cancer therapy.
11. Medically apparent CNS lymphoma or leptomeningeal disease.
12. Current or previous history of CNS disease.
13. Major surgery or significant traumatic injury < 28 days prior to the first dose of the study drug.
14. Patients with another invasive malignancy in the last 2 years.
15. Significant cardiovascular disease or active pulmonary disease.
16. Received systemic immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 Dose Escalation：The maximum tolerated dose (MTD) | Incidence of dose limiting toxicities (DLTs) up to 28 days
  To determine the maximum tolerated dose (MTD)
Part 2 Dose Expansion：ORR | Up to 2 years
  To assess anti-tumor activity of Orelabrutinib (ICP-022) in Patients with B-cell malignancies including r/r MCL, r/r FL, r/r MZL and CLL/SLL with/without prior treatment.

SECONDARY OUTCOMES:
Part 1 Dose Escalation：Incidence and severity of treatment-emergent adverse events (AEs) [Safety and Tolerability] | Up to 2 years
  The incidence and severity of treatment-emergent AEs will be collected and the safety and tolerability of ICP-022 will be assessed
Part 1 Dose Escalation：ORR | Up to 2 years
  Objective response rate
Part 1 Dose Escalation：T1/2 | Up to 2 years
  Elimination half-life
Part 2 Dose Expansion：Incidence and severity of treatment-emergent adverse events (AEs) [Safety and Tolerability] | Up to 2 years
  The incidence and severity of treatment-emergent AEs will be collected and the safety and tolerability of ICP-022 will be assessed
Part 2 Dose Expansion：DOR | Up to 2 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (36):
- United States (27):
  - Mayo Clinic-Mayo Clinic Hospital-Phoenix, Phoenix, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - Los Angeles Cancer Network - Good Samaritan Hospital Location, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - The Oncology Institute of Hope & Innovation, Whittier, California
  - Florida Cancer Specialists (FCS) South, Fort Myers, Florida
  - Asclepes Research Centers - Weeki Wachee, Weeki Wachee, Florida
  - Northwest Neurology - Rolling Meadows Office, Elk Grove Village, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Cotton O'Neil Cancer Center (Stormont-Vail Cancer Center), Topeka, Kansas
  - Tulane University School of Medicine - Tulane Cancer Center Comprehensive Clinic TCCCC, New Orleans, Louisiana
  - Anne Arundel Medical Center (AAMC) Oncology and Hematology, Annapolis, Maryland
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Summit Medical Group, Florham Park, New Jersey
  - Clinical Research Alliance, Westbury, New York
  - Gabrail Cancer Research Center, Canton, Ohio
  - University of Pittsburgh - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Cancer Center, Sayre, Pennsylvania
  - Prairie Lakes Cancer Center, Watertown, South Dakota
  - Tennessee Oncology - Chattanooga Oncology & Hematology Associates, Chattanooga, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Medical Oncology Associates PS (dba Summit Cancer Centers), Spokane, Washington
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Carmel Medical Center, Haifa
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- Ukraine (6):
  - Cherkassy Regional Oncology Center, Cherkasy
  - Khmelnytskyi Regional Hospital, Khmelnytskyi
  - St. Luke's Hospital - Medical and Diagnostic Center, Kropyvnytskyi
  - National Cancer Institute, Kyiv
  - Institute of Blood Pathology and Transfusion Medicine, Lviv
  - Transcarpathian Regional Clinical Hospital named after Andrii Novak, Uzhhorod